CLINICAL TRIAL: NCT00135733
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study of the Efficacy and Safety of Alefacept in the Treatment of Moderate to Severe Erosive Mucosal Lichen Planus
Brief Title: A Safety and Efficacy Study of Alefacept in the Treatment of Moderate to Severe Erosive Mucosal Lichen Planus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical sponsor withdrew financial support.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Stanford University (Other); Biogen (Industry)
Responsible Party: Alexandra Kimball, MD, MPH, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004P002141
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Lichen Planus
Keywords: Lichen Planus; Mucosal lichen planus; Alefacept; T-cell mediated; subcutaneous medication; Autoimmune disease
MeSH Terms: conditions — Lichen Planus; Autoimmune Diseases | interventions — Alefacept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Amevive
  Interventions: Drug: Amevive (Alefacept)
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amevive (Alefacept)
  Arms: A
Drug: Placebo
  Arms: B

SUMMARY:
The purpose of this study is to find out how safe and effective an investigational drug called alefacept (amevive) is for the treatment of moderate to severe erosive mucosal lichen planus.

Lichen planus is a skin disease that can last a long time and cause significant pain, itching, and scarring. It can affect the mucous membranes (area inside the mouth and vagina) and these areas can become erosive (sores can develop). Currently there is no known cure for this disease.

An investigational drug is one that has not been approved by the United States (US) Food and Drug Administration (FDA) to treat a particular condition or disease. Alefacept has been approved to treat psoriasis (a scaly skin rash). A number of reports suggest that lichen planus develops for some of the same reasons as psoriasis, but alefacept is not yet approved for the treatment of psoriasis.

DETAILED DESCRIPTION:
Lichen planus is an inflammatory disorder that affects skin, mucous membranes (the skin in the mouth and vagina), nails, and hair. It is thought that T-cells (cells that help fight infection) become activated and multiply faster than normal and that this contributes to the development of the skin sores.

Alefacept works by slowing the rate at which T-cells become activated and helps to decrease the number of T-cells. By blocking the activity and decreasing the number of T-cells Alefacept may help improve the disease and decrease the sores on the skin.

Participants in this study will be randomly assigned to receive either alefacept or a placebo. A placebo looks just like the study drug but contains no active medication. Placebos help study doctors find out if the effects of the study drug are due to the drug itself or just because of being in the study. This type of study design helps measure the true effectiveness of a treatment. Participants have a 1 out of 2 chance of receiving alefacept and a 1 out of 2 chance of receiving placebo. Neither participants nor the study doctors will know which group participants have been assigned to.

The researchers expect to enroll 26 subjects in this study at research sites in the U.S. About 16 subjects will be enrolled at Brigham and Women's Hospital and Massachusetts General Hospital.

Biogen Idec., Inc. is the maker of alefacept and is the sponsor of this study.

If taking part in another research study or have taken part in a research study in the last 28 days, individuals will not be able to take part in this study. Patients cannot be on multiple studies simultaneously; however, exceptions are made for non-invasive, non-interventional, and observational studies.

This study will last 24 weeks, with a total of 16 visits; screening week 0 (baseline), weeks 1-12, week 16 and week 24. Participants will not be allowed to use any oral or injectable medications for lichen planus during this study. Participants also will not be allowed to use certain creams for lichen planus during the study. The study consists of weekly injections of the medication for 12 weeks and then a 12 week follow up period.

All participants must be at least 18 years of age with a diagnosis of moderate to severe mucosal lichen planus. Neither pregnant nor nursing women will be included in the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent, authorize release and use of protected health information
* At least 18 years of age
* Diagnosis of moderate to severe mucosal lichen planus
* No systemic (oral or injectable) treatment of lichen planus for 4 weeks prior to starting study drug.
* Willing to forgo changes in topical treatment (creams) for 4 weeks before receiving the study drug and during the course of the study.
* Off of topical tacrolimus or pimecrolimus for 4 weeks prior to starting the study drug
* CD4+ T lymphocyte counts must be above the lower limit of normal laboratory value

Key Exclusion Criteria:

* Clinically significant abnormal laboratory values
* Skin lesions currently undiagnosed, but suspicious for malignancy
* Other skin disease that might interfere with lichen planus status assessments.
* History of malignancy other than basal cell carcinomas or fewer than 3 squamous cell carcinomas
* Exposure to systemic therapy for lichen planus within 4 weeks prior to enrollment.
* Previous exposure to alefacept

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Statistically significant changes in pain level
Statistically significant changes in appearance of lesions (sores)

SECONDARY OUTCOMES:
Statistically significant changes in severity of itching
Statistically significant changes in redness, amount of body surface area involved, number of sores, and or depth of involvement
Statistically significant changes in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B. Kimball, MD, MPH, Principal Investigator — CURTIS - Clinical Unit for Research Trials in Skin at Partners (MGH and BWH)
Locations (1):
- Clinical Unit for Research Trials in Skin, Boston, Massachusetts, United States

REFERENCES:
- [Background] Daoud MS, Pittelkow MR, Fitzpatrick's Dermatology in General Medicine, sixth edition, ed. Freedberg IM, Eisen AZ, Wolff K, Austen KF, Goldsmith LA, Katz SI, McGraw-Hill, pp 463-476, 2003.
- [Background] Stewart EG, Vulvar Lichen Planus, Up To Date, version 12.3, Aug 2004.